CLINICAL TRIAL: NCT07118540
Title: Evaluation of the Care Provided to Patients Who Underwent Bariatric Surgery and Were Lost to Follow-up 5 Years After Surgery
Acronym: OBEPER
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NOMINE-CRIQUI Claire, Staff surgeon in Visceral Metabolic and oncologic surgery department, head of the endocrine surgery Unit, Central Hospital, Nancy, France
Other Study IDs: 16062025
Record Dates: First submitted 2025-07-08; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
Keywords: obesity; bariatric surgery; overweight; lost to follow-up
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2025, bariatric surgery combined with nutritional and psychological support is one of the most effective treatments for patients with morbid obesity. (2)(3)

However, it causes various deficiencies, such as vitamin and iron deficiencies, which justify lifelong personalised vitamin supplementation and, consequently, lifelong medical supervision. The latest recommendations from the French National Authority for Health (Haute Autorité de Santé) clearly state that patients must commit to lifelong medical follow-up after bariatric surgery. (HAS, February 2024, R94). R94. Regular biological monitoring after bariatric surgery is recommended: three times in the first year and then once or twice a year thereafter.

Within the OBESEPI cohort (clinical trial number NCT02663388), which comprises patients who underwent surgery at Nancy University Hospital between 2013 and 2018, we observed that over 50% of patients were lost to follow-up five years after surgery.

DETAILED DESCRIPTION:
Duration of the inclusion period: 3 months Duration of subject participation (from inclusion to the last visit for the same subject): 30 minutes (time required to complete the questionnaire) Total duration of the research: 9 months

Patients with obesity who met the HAS (French high health authority) criteria for surgical treatment were recruited.

This corresponds to patients with a BMI > 35 kg/m2 with obesity-related complications (hypertension and/or diabetes and/or dyslipidemia and/or obstructive apnea syndrom ) and patients with a BMI > 40 with or without obesity-related complications.

These patients, who were candidates for scheduled bariatric surgery, were recruited by a surgeon involved in the protocol during preoperative consultations in the Metabolic, Visceral and oncologic department of surgery ; Department at Nancy University Hospital; between 2013 and 2018 (the OBESEPI-ALDEPI cohort - clinical trial NCT02663388) ). All patients met the HAS's eligibility criteria previously cited for bariatric surgery.

Two groups could be studied:

Patients who underwent surgery and were lost to follow-up five years after after bariatric surgery

The second group comprised patients who underwent surgery and were still being monitored at Nancy University Hospital five years after their inclusion.

Patients were considered lost to follow-up if there was no record of them visiting the Metabolic, Visceral and oncologic department of surgery five years after their inclusion, as determined using the DXCare software (which contain medical file).

A questionnaire is used to collect all data. This is completed by telephone or sent by email to patients who have been lost to follow-up.

This questionnaire contains questions designed to help us achieve the main and secondary objectives described in the dedicated section.

Statistical analysis :

All data will be presented as numbers and percentages for qualitative variables, and as means, standard deviations, medians, quartiles, and extreme values for quantitative variables.

The characteristics of patients lost to follow-up from the OBESPI cohort will be compared with those still being followed up using Fisher's exact test, Chi-squared test or Wilcoxon's rank sum test.

To meet the objectives, these tests will also be used to compare patients lost to follow-up with those still being followed.

Assessment of research benefits:

Methods for monitoring patients lost to follow-up should be assessed in order to develop training for general practitioners in the Lorraine region, enabling them to provide appropriate follow-up care to patients who have undergone bariatric surgery.

Train general practitioners to prevent nutritional complications of bariatric surgery.

Train general practitioners to recognise the warning signs that require referral to a specialist centre.

There is major interest in improving healthcare practices, given that 60,000 bariatric surgeries are performed annually in France, with 800,000 patients having undergone surgery in 2019.

ELIGIBILITY:
Inclusion Criteria:

* > Patients included in the OBESEPI cohort;

  * Individuals who have received complete information about the organisation of the research and have not objected to their participation and the use of their data;
  * Affiliation with a social security scheme.

Exclusion Criteria:

* >Patient who objects to participating in this research;

  * Pregnant and breastfeeding women;
  * Patients under legal guardianship or curatorship;
  * Patients deprived of their liberty by a judicial or administrative decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients were obese with BMI> 35kg/m2. These patients, who were candidates for scheduled bariatric surgery, were recruited during preoperative consultations by surgeons involved in the protocol at the Digestive, Hepatobiliary, Endocrine and Oncology Surgery Department at Nancy University Hospital between 2013 and 2018 (the OBESEPI cohort).
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Assess the proportion of patients lost to follow-up from the OBESEPI cohort who are still receiving medical care (at another centre or from their general practitioner)in %. | from bariatric surgery to 5 years after
  Assess the proportion of patients lost to follow-up from the OBESEPI cohort who are still receiving medical care (at another centre or from their general practitioner) in %.

SECONDARY OUTCOMES:
Describe the reasons for discontinuing post-bariatric surgery follow-up at Nancy University Hospital. | from surgery to 5 years after
  1.Describe the reasons for discontinuing post-bariatric surgery follow-up at Nancy University Hospital using a questionnaire :
  * I am doing well (%)
  * I do not see the point (%)
  * I live far away (%)
  * I do not have time (%)
  * other reason (%)
Describe how often patients lost to follow-up by Nancy University Hospital are followed up by another centre or their attending physician | from surgery to 5 years after
  Describe who follow the patients lost to follow-up by the referral center :
  * another center (%)
  * their attending physician (%)
  * no follow-up for bariatric surgery
Compare the proportion of patients receiving vitamin supplementation between those lost to follow-up in the OBESEPI cohort and those still being monitored. | from time of surgery to 5 years after
  Compare the proportion of patients receiving vitamin supplementation between those lost to follow-up in the OBESEPI cohort and those still being monitored.
  * % of patient who received Vitamin D in the 2 groups
  * % of patients who received vitamin B12 in the 2 groups
  * % of patients who received zinc in the 2 groups
Compare comorbidities in patients lost to follow-up in the OBESEPI cohort with those in patients still being monitored (in %) | from surgery to 5 years after
  Compare comorbidities of obesity frequency between patients lost to follow-up and patients still being monitored :
  * hypertension (%),
  * diabetes (%),
  * dyslipidaemia (%)
  * obstructive sleep apnoea ( %)
Compare the proportion of post-bariatric surgery complications requiring surgery (%) | from bariatric surgery to 5 years after
  Compare the proportion of post-bariatric surgery complications requiring surgical intervention among the groups 2 groups (patients lost to follow up compared to patients who are still being monitored) (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] (1)Global, regional, and national prevalence of adult overweight and obesity, 1990-2021, with forecasts to 2050: a forecasting study for the Global Burden of Disease Study 2021 Lancet. 2025 Mar 8; (2)Peirson L, Douketis J, Ciliska D, Fitzpatrick-Lewis D, Ali MU, Raina P. Treatment for overweight and obesity in adult populations: a systematic review and meta-analysis. CMAJ Open. Oct 2014;2(4):E306-317. (3)Jackson VM, Breen DM, Fortin JP, et al. Latest approaches for the treatment of obesity. Expert opinion on drug discovery. 2015;10(8):825-839. (4)Recommandation HAS février 2024 : Prise en charge de l'obésité de niveau 2 et 3 https://www.has-sante.fr/upload/docs/application/pdf/2024-02/reco369_recommandations_obesite_2e_3e_niveaux_ii_cd_2024_02_08_preparation_mel.pdf (5)Chirurgie bariatrique : état des lieux en France en 2019 Halimi et al Médecine des maladies Métaboliques